CLINICAL TRIAL: NCT00341302
Title: A Prospective, Observational Study of HIV-Infected Pregnant Women and HIV-Exposed, Uninfected Children at Clinical Sites in Latin American Countries
Brief Title: A Prospective, Observational Study of HIV-Infected Pregnant Women and Their Infants at Clinical Sites in Latin American and Caribbean Countries
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902261; 02-CH-N261
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Pregnant HIV Positive Women
Keywords: HIV; AIDS; Perinatal; Transmission; Outcomes
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Cohort 1: HIV Infected Pregnant Women
- Pediatric Cohort 2: HIV exposed , uninfected children born to HIV infected women
- Pediatric Cohort 3: HIV exposed, uninfected children 6 months to 5 years of age

SUMMARY:
By the end of 1999, it was estimated that 1.2 million children were living with HIV infection. During 1999 alone, 600,000 children were newly infected with HIV, mostly in less-developed countries. Most HIV-infected children are infected by transmission from mother to child during pregnancy, at birth, or through breast milk. Antiretroviral medications, cesarean section before rupture of membranes, and avoidance of breastfeeding are ways to reduce the risk of transmission. This study will determine mother-to-child transmission rates and the effects on infants of exposure to antiretroviral medications and mode of delivery.

Approximately 180 to 240 HIV-infected pregnant women in Mexico and Argentina will be enrolled during the first year of this 5-year study. HIV-infected women will be evaluated during pregnancy, during delivery, and 6 months after delivery. At each visit, a history will be taken and physical examination given; blood will be collected for laboratory tests.

HIV-exposed infants will be evaluated through 6 months of age. At each of 2 visits, a history will be taken and physical examination given; blood will be collected for laboratory tests; and growth will be assessed.

DETAILED DESCRIPTION:
This is an observational, prospective cohort study to describe the characteristics of HIV-infected pregnant women and HIV-exposed, uninfected children at participating clinical sites in Latin America where the following are available: 1) antiretrovirals (ARVs) for treatment of HIV-infected women and for prevention of mother-to-child transmission (MTCT) of HIV; and 2) infant formula. We will describe the utilization of interventions related to decreasing the risk of MTCT, including ARV prophylaxis, cesarean section before labor and before ruptured membranes, and complete avoidance of breastfeeding. We will describe receipt of maternal ARV regimens and determine rates of MTCT of HIV. This study will describe maternal adverse events during pregnancy and the postpartum period. In addition, the study will describe child outcomes potentially related to in utero and early postnatal exposure to ARVs. HIV-infected women will be evaluated antepartum, intrapartum, 6 months postpartum and then every 6 months for up to 5 years after delivery. HIV-exposed, uninfected children will be evaluated for up to 5 years of follow-up.

ELIGIBILITY:
* INCLUSION CRITERIA: (HIV-Infected Pregnant Women)

Pregnant women at 22 weeks of gestation or more with documentation of pregnancy, using one or more of the following:

Urine HCG pregnancy test;

Serum HCG pregnancy test;

Positive fetal heart tones by Doppler; or

Ultrasound.

Documentation of HIV infection, defined by any two of the following prior to or during pregnancy:

Reactive test for HIV antibody;

Positive HIV culture;

Positive HIV DNA PCR;

Positive neutralizable HIV p24 antigen;

Positive qualitative HIV RNA;

Quantitative HIV RNA greater than or equal to 1000 copies/ml; and

Diagnosis of AIDS-defining clinical condition.

Willingness and intent to deliver at the participating clinical site and to be followed through six months postpartum at the site or associated outpatient facility.

Willingness and ability to sign informed consent-Subject must be of an age to provide legal informed consent as defined by the country in which the subject resides.

Willingness and intent to have children followed for up to 5 years.

Subjects may be co-enrolled in clinical trials for treatment or prophylaxis of HIV infection, opportunistic infections, or other HIV related problems.

Subjects may be re-enrolled with subsequent pregnancies during this study. However, if so, their follow-up for the previous pregnancy will be discontinued. Children from each pregnancy will be followed in accordance with the protocol.

Subjects may enroll up to and prior to delivery, including during labor.

INCLUSION CRITERIA: (Dynamic Pediatric Cohort)

-HIV-exposed children born to enrolled HIV-infected pregnant women. Children diagnosed with HIV infection will be discontinued from the present protocol and(if eligible) offered enrollment into a concurrent NICHD-funded protocol for HIV-infected children.

INCLUSION CRITERIA: (Static Pediatric Cohort)

-HIV-exposed, uninfected children who are 6 months of age through 5 years 364 days of age and were previously enrolled in the NISDI Pediatric Protocol or NISDI Perinatal Protocol.

And

* Other HIV-exposed, uninfected children who are 6 months of age through 5 years 364 days of age at time of enrollment into this protocol.

  1. Documentation of HIV-uninfected status should be obtained from medical

     record review.
  2. Evidence of the HIV-uninfected status of the infants and children can be documented by the following:

     --Two or more negative HIV virologic assays (e.g., HIV culture or HIV DNA PCR) with one test performed at age 1 month or older and one performed at age 4 months or older, and no positive virologic tests.

     Or

     --One or more negative HIV virologic assays performed at 1 month of age or older with one or more negative HIV antibody tests (including HIV rapid tests) performed at greater than or equal to 6 months of age.

     Or

     --One positive HIV virologic assay, with at least two later negative HIV virologic tests (at least one of which is after age 4 months of age) or negative HIV antibody tests (at least one of which is after 6 months of age).
  3. Documentation of HIV infection in the mother must have been obtained either prior to or during pregnancy or within one month postpartum.
  4. Evidence of HIV infection in the mother can be documented by two or more of the following:

     * Reactive test for HIV antibody;
     * Positive HIV culture;
     * Positive HIV DNA PCR;
     * Positive quantitative HIV p24 antigen above assay cutoff;
     * Positive qualitative HIV RNA;
     * Quantitative HIV RNA >= 1000 copies/ml; and
     * Diagnosis of AIDS-defining clinical condition.
  5. Complete data regarding maternal medications received during pregnancy must be available through medical record abstraction.

     EXCLUSION CRITERIA: (HIV-Infected Pregnant Women)

     Failure to meet inclusion criteria.

     EXCLUSION CRITERIA: (Dynamic Pediatric Cohort)
* Failure to meet inclusion criteria

EXCLUSION CRITERIA: (Static Pediatric Cohort)

* HIV infection of the child
* Insufficient documentation of HIV infection in the mother obtained either prior to or during pregnancy or within one month postpartum.
* Insufficient evidence of HIV infection in the mother
* Insufficient perinatal data

  1. Incomplete data regarding maternal medications received during pregnancy (e.g., missing start and stop dates).
  2. Incomplete data regarding postnatal ARV exposure.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV -infected pregnant women and HIV exposed, uninfected children followed at participating Latin American sites@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 3554 (Actual)
Dates: Start 2002-07-25 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
To describe the characteristics of HIV-infected pregnant women and their HIV-exposed children in Latin America, including the rates of and risk factors for mother-to-child transmission | in utero, six weeks
  To describe the characteristics of HIV-infected pregnant women and their HIV-exposed children in Latin America, including the rates of and risk factors for mother-to-child transmission.
To characterize adverse events according to receipt of and exposure to ARVs (by HIV- infected women during pregnancy and postpartum and by their HIV-exposed but uninfected children in utero and during the first few week | in utero, six weeks
  To characterize adverse events according to receipt of and exposure to ARVs (by HIV- infected women during pregnancy and postpartum and by their HIV-exposed but uninfected children in utero and during the first few week

CONTACTS AND LOCATIONS:
Overall Officials: Nahida A Chakhtoura, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (12):
- Hospital General de Agudos "Jose Maria Ramos Mejia", Buenos Aires, Argentina
- Brazil (10):
  - Universidade de Caxias do Sul, Caxias do Sul
  - Universidade Federal de Minas Gerais, Minas Gerais
  - Hospital Geral Nova de Iguacu Setor De DST/AIDS, Nova Iguaçu
  - Hospital Conceicao, Porto Alegre
  - Hospital Femina, Porto Alegre
  - Irmandade Da Santa Casa de Misericordia de, Porto Alegre
  - Hospital dos Servidores do Estado - RJ, Rio de Janeiro
  - Instituto de Puericultura e Pediatria, Rio de Janeiro
  - Federal University of Sao Paulo-Escola Paulista de Medicina, São Paulo
  - Hospital das Clinicas da Falculdade De Medinica, São Paulo
- Unversity of San Marcos, Lima, Peru

REFERENCES:
- [Background] Rates of mother-to-child transmission of HIV-1 in Africa, America, and Europe: results from 13 perinatal studies. The Working Group on Mother-To-Child Transmission of HIV. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Apr 15;8(5):506-10. doi: 10.1097/00042560-199504120-00011. PMID 7697448
- [Background] U.S. Public Health Service recommendations for human immunodeficiency virus counseling and voluntary testing for pregnant women. MMWR Recomm Rep. 1995 Jul 7;44(RR-7):1-15. PMID 7565546
- [Background] Connor EM, Sperling RS, Gelber R, Kiselev P, Scott G, O'Sullivan MJ, VanDyke R, Bey M, Shearer W, Jacobson RL, et al. Reduction of maternal-infant transmission of human immunodeficiency virus type 1 with zidovudine treatment. Pediatric AIDS Clinical Trials Group Protocol 076 Study Group. N Engl J Med. 1994 Nov 3;331(18):1173-80. doi: 10.1056/NEJM199411033311801. PMID 7935654